CLINICAL TRIAL: NCT06716086
Title: A Novel Shape Memory Alloy-Based Orthosis for Proximal Interphalangeal Joint Stiffness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-113-251
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Finger Proximal Interphalangeal Joint Contracture
Keywords: shape memory alloy; finger stiffness; joint contracture; joint range of motion; hand injury
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMA group (Experimental): Participants in the SMA group will use the shape memory alloy-based orthosis. They will undergo a 30-minute home-based training program 3-4 times a day, 7 days a week, for 8 weeks.
  Interventions: Other: shape memory alloy-based orthosis
- Stretching group (Active Comparator): Participants in the Stretching group will receive conventional stretching program as a home program. They will undergo a 30-minute home-based training program 3-4 times a day, 7 days a week, for 8 weeks.
  Interventions: Other: conventional stretching program

INTERVENTIONS:
Other: shape memory alloy-based orthosis — The home program with the shape memory alloy-based orthosis contains warm-up part and correction part. The SMA-based orthosis is an improvement over traditional dynamic splint. This corrective device uses shape memory alloy as an elastic component specifically designed to address finger joint stiffness. It provides continuous force for stiff joint in order to address stiffness.
  Arms: SMA group
Other: conventional stretching program — The home program for the stretching group includes active joint range of motion exercises and passive stretching exercises. Participants will follow instructions to perform various joint movements, with a focus on their restricted fingers.
  Arms: Stretching group

SUMMARY:
The goal of this clinical trial is to evaluate the applicability, effectiveness, and usability of a shape memory alloy-based orthosis for patients with finger proximal interphalangeal joint stiffness. This cutting-edge design incorporates shape memory alloy into the device for improving proximal interphalangeal joint stiffness and, secondarily, enhancing the ability to perform activities.

Half of the participants will be assigned to experimental group, receiving a shape memory alloy-based orthosis for home program. The other half will be assigned to control group, receiving a conventional stretching program. Three evaluations, examining range of motion and hand functional performance, will be conducted before intervention, 4 weeks and 8 weeks after baseline by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years old
* Exhibit limitations in passive range of motion of the proximal interphalangeal joint, with extension less than 0 degrees or flexion less than 90 degrees.
* Beyond the acute phase of the hand condition, and it has been more than 8 weeks post-surgery (or post-injury).

Exclusion Criteria:

* Concurrently use other types of splints for PIP joint stiffness.
* Present with abnormal muscle tone, paralysis, or rigidity associated with central or peripheral nervous system dysfunction.
* Suffer from complex regional pain syndrome or progressive degenerative disease affecting finger joints, such as rheumatoid arthritis.
* Have an active infection or arthritis in their fingers.
* Unable to follow instructions.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Range Of Motion | Baseline, 4 weeks after baseline, and 8 weeks after baseline
  Active, passive and torque range of motion are common measurements to assess joint mobility limitations in clinical settings. Active range of motion is measured as the maximum movement achieved by the patient's own efforts. Passive range of motion is measured when an external force, such as a therapist, moves the joint until the end feel is detected. Torque range of motion is assessed with a specific tension applied to the movement of interest. Normal proximal interphalangeal joint flexion range of motion typically ranges from 0-100 or 110 degrees.

SECONDARY OUTCOMES:
Minnesota Manual Dexterity Test | Baseline, 4 weeks after baseline, and 8 weeks after baseline
  The Minnesota Manual Dexterity Test assesses fine manual dexterity and consists of two subtests: the placing and turning tests. These involve hand movements such as picking up, turning, transferring, and placing disks. Each subtest includes two trials, resulting in a total of six trials. The combined time taken to complete both trials in each subtest will be recorded.
Purdue Pegboard Test | Baseline, 4 weeks after baseline, and 8 weeks after baseline
  The Purdue Pegboard Test assesses fine motor coordination and manipulative ability through four subtests: dominant hand, non-dominant hand, both hands, and assembly. In each subtest, participants place as many pins as possible in the designated column, with the assembly subtest also incorporating washers and collars. The allotted time is thirty seconds for the dominant hand, non-dominant hand, and both hands subtests, and sixty seconds for the assembly subtest. Each subtest is repeated three times, and the average of these three trials is calculated as the final score.
Motion Capture and Analysis System | Baseline, 4 weeks after baseline, and 8 weeks after baseline
  The motion capture system will be used to measure the functional range of motion of the hand. It utilizes standard cameras or Vicon motion capture system to record hand movements of participants. The data is further analyzed using tools such as MATLAB, Mediapipe, or other motion analysis software to assess the functional range of motion of the hand.
The Disability of the Arm, Shoulder and Hand Questionnaire, Taiwan version | Baseline, 4 weeks after baseline, and 8 weeks after baseline
  The Taiwan version of the Disability of the Arm, Shoulder, and Hand Questionnaire is a 30-item, self-reported tool used to assess hand function, specifically addressing physical function and symptoms in patients with upper limb musculoskeletal disorders. It provides a detailed view of patient disability and tracks changes in symptoms and function over time. Each item is scored on a 5-point Likert scale, where 1 represents no difficulty and 5 represents inability to perform the task. Responses are based on the patient's experiences from the past week, with scores converted to a 0-100 scale, where higher scores indicate greater severity of disability.
System Usability Scale | 8 weeks after baseline
  The System Usability Scale assesses the usability of the SMA-based orthosis. It evaluates effectiveness and satisfaction from the user's subjective perspective. The scale contains 10 items, each with five response options, where 1 means "Strongly disagree" and 5 means "Strongly agree". Participants' scores for each item are converted to range from 0 to 4. For items 1,3,5,7, and 9, the converted score is the participant's scores minus 1. For items 2,4,6,8 and 10, the converted score is 5 minus the participant's scores. The sum of these scores is then multiplied by 2.5 to obtain the overall usability value.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No